CLINICAL TRIAL: NCT02802696
Title: Pre-transfusion Furosemide in Patients at High Risk of Transfusion-associated Circulatory Overload - The Transfusion-Associated Circulatory Overload Best Eliminated With Lasix (TACO-BEL) Study: A Pilot Randomized Controlled Trial
Brief Title: Transfusion-Associated Circulatory Overload Best Eliminated With Lasix
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University Health Network, Toronto (Other); Canadian Blood Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16-5032
Record Dates: First submitted 2016-02-29; First posted 2016-06-16 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2016-10

CONDITIONS: Transfusion-associated Circulatory Overload
Keywords: Transfusion; Transfusion Medicine; Diuretic
MeSH Terms: conditions — Transfusion Reaction | interventions — Furosemide; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Furosemide (Experimental): Diuretic
  Interventions: Drug: Furosemide
- Placebo (Placebo Comparator): Normal saline
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Furosemide — A bolus dose of 20mg furosemide (20mg/2mL) will be given intravenously by slow intravenous push within 60 minutes prior to the start of the red blood cell transfusion; infusion via minibag is also acceptable.
  Other Names: Lasix
  Arms: Furosemide
Drug: Normal Saline — A single bolus dose of 2 mL normal saline will be given intravenously immediately within 60 minutes prior to the start of the red blood cell transfusion; infusion via minibag is also acceptable.
  Other Names: 0.9% Sodium Chloride
  Arms: Placebo

SUMMARY:
This is a pilot double-blinded placebo-controlled randomized controlled trial (RCT) to evaluate the feasibility of conducting a multicenter, randomized, placebo-controlled trial to assess the efficacy of pre-transfusion furosemide in preventing transfusion-associated circulatory overload (TACO) in hemodynamically stable inpatients aged 65 years or older receiving a single unit red blood cell transfusion. Patients will be randomly allocated to receive either furosemide (20mg intravenous) or placebo (saline) within 60 minutes of starting a red blood cell (RBC) transfusion. Randomization will be stratified by centre and renal dysfunction (creatinine clearance ≥ 60 mL/min or < 60 mL/min). This is a blinded trial: patients, care-providers (physicians and nurses), data collectors, outcome adjudicators, and data analysts will not be aware of group allocation.

DETAILED DESCRIPTION:
The investigators proposed this pilot study to assist us in determining the feasibility of conducting a definitive multicenter randomized trial across Canada.

Rationale:

The rationale for this study includes: (1) TACO is the leading cause of morbidity and mortality due to transfusion; (2) risk factors for TACO include older age, renal dysfunction and positive fluid balance; (3) furosemide is a diuretic commonly prescribed for fluid overload; (4) furosemide can decrease pulmonary artery pressures; and (5) clinical uncertainty as to the effect of furosemide in preventing TACO. The investigators will enroll 80 patients in this pilot study at two centers.

Hypothesis:

The investigators hypothesize that 80 patients can be enrolled in the trial within a 2-month period

Justification:

If pre-transfusion that furosemide decreases the rate of TACO with red blood cell transfusion, clinical practice worldwide would change. Over 800,000 patients in Canada receive a blood transfusion annually and many are at high risk for TACO and may benefit from this simple, low-cost intervention. This intervention could easily be generalizable worldwide. There are practical challenges related to patient recruitment, adherence to trial protocol and data collection, all of which the TACO-BEL Pilot Trial will seek to measure.

Objectives:

The primary outcome of this trial is to determine the feasibility of performing a large multi-centre, randomized, placebo-controlled trial with concealed allocation and blinded outcome assessment, adequately powered to determine a clinically significant effect of pre-transfusion furosemide on the incidence of transfusion-associated circulatory overload.

Primary outcome measure is the number of patients enrolled within a two-month period

Secondary feasibility outcome measures include:

1. Proportion of patients screened meeting eligibility criteria
2. Proportion of eligible patients consenting to participate
3. Proportion of consenting patients receiving the allocated treatment
4. Proportion of treated patients completing follow-up assessment
5. Proportion of patients in which blinding was maintained throughout study

Research Method:

Patients meeting inclusion criteria will be identified by reviewing transfusion orders received by the blood transfusion laboratory or by referral from ordering physicians; these patients will then be approached by study personnel to obtain pre-transfusion informed consent. Randomization will be performed by pharmacy at the time of drug preparation. The randomization code will be generated in random blocks of 4 to 6, stratified by center, and renal function at time of randomization (creatinine clearance < 60 and ≥ 60 mL/min) using a computer based randomization program.

Intervention:

Patients will be administered a bolus dose of 20mg furosemide (20mg/2mL) intravenously within 60 minutes prior to the start of the red blood cell transfusion. Patients randomized to placebo will be administered an equal volume of normal saline intravenously immediately within 60 minutes prior to the start of the red blood cell transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years.
* Receiving a single unit red blood cell transfusion

Exclusion Criteria:

* Active bleeding (active visible bleeding, required 2 or more RBC units in the preceding 24 hours, drop in Hb > 20 g/L in the preceding 24 hours);
* Hemodynamically unstable (systolic blood pressure < 90 mmHg or on inotropes);
* Anticipated major surgical procedure within 24 hours of enrolment;
* Presence of hyponatremia (Na < 130 mmol/L);
* Presence of hypokalemia (K < 3.5 mmol/L);
* Dialysis or creatinine clearance < 30 mL/min;
* Order for platelet or plasma transfusion at same time;
* Allergy to furosemide;
* Risk of withholding furosemide felt by attending physician to place patient at excessive risk of harm;
* Previously enrolled in the study;
* Plan for discharge on the day of randomization;
* Unable to provide informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-06; Primary Completion 2017-03-17 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
Number of patients enrolled | 2 months period

SECONDARY OUTCOMES:
Proportion of patients screened meeting eligibility criteria | 2 months
Proportion of eligible patients consenting to participate | 2 months
Proportion of patient receiving the allocated treatment | 2 months
Proportion of treated patients completing follow-up assessment | 2 months
Proportion of patient in which blinding was maintained throughout study | 2 months
Vital Signs | Baseline and 6 hours post transfusion
  Change in vital signs immediately post-transfusion and at 6 hours post-transfusion
Positive end-expiratory pressure | Baseline and 6 hours post transfusion
  For patients on mechanical ventilation pre-transfusion, change in positive end-expiratory pressure
Inspiratory oxygen | Baseline and 6 hours post transfusion
  change in fraction of inspiratory oxygen at 6 hours post-transfusion
Incidence of TACO within 6 hours from completion of transfusion | within 6 hours
Severity of TACO-graded as per the Public Health Agency of Canada's Transfusion Transmitted Injuries Surveillance System | within 6 hours
Validation of TACO as per criteria adopted from the US Center for Disease Control | within 6 hours
Change in plasma brain natriuretic peptide(BNP) | Baseline and Day 1
Net fluid balance at 24 hours from start of transfusion- all intravenously-administered fluids (including the transfused blood product and the study intervention) | Within 24 hours
Proportion of patients developing hyponatremia or hypokalemia by Day 1 | By Day 1
Proportion of patients developing hypotension | Within 24 hours
Proportion of patients developing acute kidney injury | Within 24 hours
Need for increased supplemental oxygen is defined as any increase in oxygen flow ≥ 1 L/hr or (fraction of inspired oxygen)FiO2 ≥ 5% of 1 hour duration or longer, prompted by either patient symptoms or a fall in oxygen saturation(SpO2) ≥ 5% | Within 24 hours
Need for inotropic support is defined as the initiation of a continuous infusion of dopamine, dobutamine, epinephrine, or norepinephrine | Within 24 hours
Need for additional diuretic or vasodilatory therapy is defined by the prescription of non-study furosemide, hydrochlorothiazide, metolazone, or either transdermal or intravenous nitroglycerin | Within 24 hours
Occurrence of acute coronary syndrome or new arrhythmia | within 7 days
Mortality during hospital stay | Upto 30 days
Length of hospital stay | From date of admission until the date discharge from an acute care hospital or date of death from any cause, whichever came first, assessed up to 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Jeannie Callum, MD, Principal Investigator — Sunny Brook Health Sciences Centre
Locations (3):
- Canada (3):
  - Canadian Blood Services, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] AABB (2015) AABB Association Bulletin #15-02: Transfusion Associated Circulatory Overload (12/28/15). Vol. 2016,
- [Background] Alam A, Lin Y, Lima A, Hansen M, Callum JL. The prevention of transfusion-associated circulatory overload. Transfus Med Rev. 2013 Apr;27(2):105-12. doi: 10.1016/j.tmrv.2013.02.001. Epub 2013 Mar 1. PMID 23465703
- [Background] Lieberman L, Maskens C, Cserti-Gazdewich C, Hansen M, Lin Y, Pendergrast J, Yi QL, Callum J. A retrospective review of patient factors, transfusion practices, and outcomes in patients with transfusion-associated circulatory overload. Transfus Med Rev. 2013 Oct;27(4):206-12. doi: 10.1016/j.tmrv.2013.07.002. Epub 2013 Sep 26. PMID 24075097
- [Background] Sarai M, Tejani AM. Loop diuretics for patients receiving blood transfusions. Cochrane Database Syst Rev. 2015 Feb 16;2015(2):CD010138. doi: 10.1002/14651858.CD010138.pub2. PMID 25685898